CLINICAL TRIAL: NCT03064217
Title: The Use of Intraoral Imaging at Clinical Crown Lengthening Procedures
Brief Title: Intraoral Imaging at Clinical Crown Lengthening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Se-Lim Oh, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00073913
Record Dates: First submitted 2017-02-17; First posted 2017-02-24 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Dental Caries of Root Surface; Surgery
Keywords: Clinical crown lengthening; intraoral imaging; Emax crown
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Making impression at surgery (Experimental): Making impression at surgery
  Interventions: Device: Making impression at surgery
- Making impression 8 weeks after surgery (No Intervention): Making impression 8 weeks after surgery

INTERVENTIONS:
Device: Making impression at surgery — Making impression at surgery
  Arms: Making impression at surgery

SUMMARY:
Crown lengthening surgery is done when a tooth needs to be fixed with a crown. Sometimes, not enough of the tooth sticks out above the gum to support a crown. This can happen when a tooth breaks off at the gum line, or when a crown or filling falls out of a tooth and there is decay underneath. To place a crown, the dentist needs to expose more of the tooth. This is done by removing some gum tissue or bone.

After surgery, the area will heal in about three months. Then, making a crown can begin. This healing period often delays the delivery a final crown. This study is investing a way to make the final impression at the surgery to expedite the delivery of a final crown.

DETAILED DESCRIPTION:
The purpose of this prospective study is to evaluate clinical and radiographic outcomes of single unsplinted fixed restorations made with digital intraoral imaging in conjunction with clinical crown lengthening procedures (CLPs) compared ones fabricated by the conventional protocol.

Specific Aim 1: To evaluate the clinical outcomes between the experimental group (the digital impression taking at clinical crown lengthening procedures) and the control group (the conventional protocol) Hypothesis: There will be no differences in clinical parameters around the teeth between the two groups.

Approach: The investigators will conduct a prospective clinical study and will compare the changes in gingival recession, the width of keratinized gingiva, and pocket depths around the teeth between the two groups.

Specific Aim 2: To evaluate the radiographic outcome between the experimental group and the control group Hypothesis: There will be no difference in crestal bone level around teeth between the two groups.

Approach: The study will investigate the difference in crestal bone level around the teeth at baseline and 12 months between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* a single-unsplinted crown needed
* the tooth must be in the area from the canine to the second molars
* a clinical crown lengthening is required to fabricate a crown

Exclusion Criteria:

* uncontrolled hypertension
* diabetes mellitus
* subjects with a history of a long-term use of corticosteroid (> 6 months)
* subjects with a history of taking oral/IV bisphosphonates within the past 2 years
* smokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Se-Lim Oh, DMD, Principal Investigator — University of Maryland School of Dentistry
Locations (2):
- United States (2):
  - Advanced General Dentistry at UMB DS, Baltimore, Maryland
  - University of Maryland School of Dentistry, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared. The results will be published.

RESULTS

PARTICIPANT FLOW:
Groups:
- Making Impression 8 Weeks After Surgery: Making the final impression 8 weeks after surgery
Period: Overall Study
Arm/Group | Making Impression at Surgery | Making Impression 8 Weeks After Surgery
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Teeth
Groups:
- Total: Total of all reporting groups
Arm/Group | Making Impression at Surgery | Making Impression 8 Weeks After Surgery | Total
Number analyzed (Participants) | 10 | 10 | 20
Number analyzed (Teeth) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 14
  >=65 years | 5 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (22) | 45.5 (16.6) | 50.6 (19.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 4 | 2 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Crestal bone loss [Mean (Standard Deviation); unit: mm] | 1.78 (0.8) | 1.14 (0.7) | 1.6 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Pocket Depth
Description: Changes in pocket depths (the distance from the gingival margin to pocket base) at 12 months from the baseline
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Making Impression at Surgery | Making Impression 8 Weeks After Surgery
Number analyzed (Participants) | 10 | 10
mm | 2.7 (1.2) | 2.4 (1.0)
Statistical Analysis 1: Comparison: Making Impression 8 Weeks After Surgery; Test type: Superiority; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Making Impression at Surgery | Making Impression 8 Weeks After Surgery
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Making Impression at Surgery (N=10) | Making Impression 8 Weeks After Surgery (N=10)
Pain (Nervous system disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT03064217/Prot_SAP_ICF_001.pdf